CLINICAL TRIAL: NCT02118701
Title: SHARED DECISION MAKING ON A 'LIFE-AND-CARE PLAN' IN LONG-TERM CARE FACILITIES
Brief Title: SHARED DECISION MAKING IN LONG-TERM CARE FACILITIES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 258883
Record Dates: First submitted 2014-04-14; First posted 2014-04-21 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2015-05

CONDITIONS: Dementia
Keywords: Shared decision making; Dementia; Long-term care; Nursing home; Care plan
MeSH Terms: conditions — Dementia

ARMS (1):
- SDM care planning (Experimental)
  Interventions: Other: Shared Decision-Making educational training

INTERVENTIONS:
Other: Shared Decision-Making educational training

SUMMARY:
Shared Decision Making (SDM) is defined as a process where healthcare professionals and patients make decisions together, using the best available evidence. SDM, as a communication and decision method, can be used also with persons suffering from dementia. Yet, SDM with persons with dementia or even with their family caregivers is not widespread.

The present research project aims to develop and evaluate an SDM framework in care planning to be implemented in long-term care facilities, in order to obtain a constantly developing care plan that focuses not only on the medical, physical, psychosocial and spiritual needs of the resident, but that considers and documents his preferences and the actions taken by caregivers to meet them.

The current project is a controlled exploratory study. Case studies that involve a triad in each case, composed by the resident with moderate or severe dementia, his family caregiver and the professional usually taking care for the resident, will be used (n=16 professionals; n=40 residents; n=40 family caregivers). Professional caregivers of two nursing homes, one located in Italy and one in the Netherlands, will receive a specific training in SDM principles and will guide the SDM interview within the triad. Primary outcome will be the proportion of residents whose preferences and needs, together with the related actions to meet them, are known, documented and satisfied in their 'life-and-care plans'. Secondary outcomes are the residents' and family caregivers' quality of life; the family caregivers' sense of competence and the healthcare professionals' job satisfaction. Semi-structured interviews and focus group interviews will be performed to assess satisfaction with the intervention and barriers and facilitators to its implementation. Assessments are performed at baseline and six months after the intervention.

We hypothesize that the use of the SDM process in care planning will increase the number of met needs and will improve the residents' and family caregivers quality of life, the family caregivers' sense of competence and the healthcare professionals' job satisfaction.

The key element of this study is that it will contribute to our knowledge about the efficacy and feasibility of an SDM framework in care planning in long-term care facilities with persons with moderate to severe dementia.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of dementia based on the Diagnostic and Statistical Manual of Mental Disorders (DSM) IV
* from moderate to severe cognitive decline (Global Deterioration Scale from 4 to 6)
* supported by a family caregiver who can be involved

Exclusion Criteria:

* unable to pronounce simple sentences

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The proportion of residents whose preferences and needs, together with the related actions to meet them, are known, documented and satisfied in their 'life-and-care plans'. | 6 months after the SDM interview

REFERENCES:
- [Derived] Mariani E, Engels Y, Koopmans R, Chattat R, Vernooij-Dassen M. Shared decision-making on a 'life-and-care plan' in long-term care facilities: research protocol. Nurs Open. 2016 Mar 6;3(3):179-187. doi: 10.1002/nop2.42. eCollection 2016 Jul. PMID 27708828